CLINICAL TRIAL: NCT06377904
Title: Clinical and Therapeutic Characteristics of Geriatric Patients Hospitalized for Heart Failure
Brief Title: Clinical and Therapeutic Characteristics of Geriatric Patients Hospitalized for Heart Failure (AGING HF Study (AGe and Heart Failure IN Geriatrics))
Acronym: AGING HF
Status: Not yet recruiting | Type: Observational
Sponsor: Gérond'if (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A02125-40
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-03

CONDITIONS: Patients Hospitalized in Geriatrics for Heart Failure; Patients Aged 75 and Over
Keywords: Heart failure; Geriatrics; AGE
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective phase: Retrospective inclusion (using data of patients who had been hospitalized between April 2020 and December 2023)
- Prospective phase: Prospective inclusion (using data of patients hospitalized between January 2024 and August 2026)

SUMMARY:
This retrospective (between April 2020 and December 2023) then prospective (between January 2024 and August 2026), non-interventional cohort study has as its main objective to evaluate the clinical and therapeutic characteristics of patients aged 75 and over hospitalized in geriatrics for heart failure and also to evaluate the clinical characteristics and triggering factor(s) of acute heart failure.

DETAILED DESCRIPTION:
Multicenter study, including patients aged 75 and over, hospitalized in geriatrics and having suffered heart failure in the geriatric wards of 3 centers. The following elements will be collected:

* Demographic data
* History (comorbidities)
* Type of heart disease
* Frailty criteria
* Clinical signs of heart failure
* Geriatric syndromes (falls, cognitive disorders, (MMSE) confusion, malnutrition, loss of autonomy (ADL, IADL), bedsores)
* Biology available (CBC, ionogram, creatinine, NT pro BNP, BHC, troponin, TSH, HBA1C)
* ECG and echocardiography data
* Treatment on admission, during stay and on discharge
* Mode of discharge and length of stay
* Follow-up at 3, 6, 9 months and one year, through telephone calls with the patient, caregiver or attending physician. Questions will cover various aspects of health and quality of life, physical activity limitations, autonomy, symptoms, anxiety, depression, as well as neurocognitive status (using adapted questions).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 75 and over Hospitalized in a geriatric ward with heart failure No oral opposition from patient

Exclusion Criteria:

* Patient under 75 years of age Patient not wishing to participate in the study Subject under guardianship/curatorship/supervision of justice

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 75 and over hospitalized in geriatrics for heart failure
Sampling Method: Non-Probability Sample
Enrollment: 810 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Evaluate the clinical and therapeutic characteristics of elderly patients hospitalized in geriatrics for heart failure | 36 months
  To Evaluate the clinical and therapeutic characteristics of elderly patients hospitalized in geriatrics for heart failure with 80% power and 5% alpha risk and expressed as a percentage.

SECONDARY OUTCOMES:
Factors associated with patients hospitalization or rehospitalization | 12 months
  Quantitative data will be described as mean ± standard deviation. Qualitative variables will be expressed as percentages Statistical differences (hospitalized and/or deceased vs. non-rehospitalized and/or non-deceased patients) will be assessed using the Mann-Whitney U-test and Student's t-test for non-parametric and parametric continuous variables, respectively. Discrete variables will be normally distributed, and by the Mann-Whitney test for those not normally distributed. Survival curves will be drawn to analyze mortality and hospitalizations. Evaluated using the χ2 or Fisher test. Differences between groups will be assessed by ANOVA for the variables